CLINICAL TRIAL: NCT03065686
Title: Identification of Genetic Factors Implicated in Orofacial Cleft Using Whole Exome Sequencing GENEPIC
Brief Title: Identification of Genetic Factors Implicated in Orofacial Cleft Using Whole Exome Sequencing
Acronym: GENEPIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2015_843_0016
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Cleft Lip and Palate
Keywords: Cleft Lip and Palate; CL/P; WES
MeSH Terms: conditions — Cleft Lip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Identification of genetic factors (Experimental): Clinical questionnaire and analysis of genetic data obtained by exome high-throughput sequencing
  Interventions: Genetic: identification of genetic factors

INTERVENTIONS:
Genetic: identification of genetic factors — Clinical questionnaire and analysis of genetic data obtained by exome high-throughput sequencing

SUMMARY:
Despite significant progress made in identification on numerous genes and gene pathways critical for craniofacial development, several approaches, ie mutation screening of specific candidates, association studies and even genome-wide scans have largely failed to reveal the molecular basis of NS human clefting

DETAILED DESCRIPTION:
Despite significant progress made in identification on numerous genes and gene pathways critical for craniofacial development, several approaches, ie mutation screening of specific candidates, association studies and even genome-wide scans have largely failed to reveal the molecular basis of NS human clefting. Moreover, the efficiency of Whole Exome Sequencing -WES- was proven. The efficiency of WES was proven by the identification of the genes causing Freeman Sheldon and Miller's syndrome, followed by several others. In the Picardy region, management and follow-up of orofacial cleft patients are well-organised by a multidisciplinary team in the university hospital of Amiens. The investigators therefore decided to perform whole exome sequencing (WES) on precisely phenotyped non-syndromic CL/P patients followed in our center.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a NSCL/P or CL/P of unknown etiology,
* national health care insurance holders

Exclusion Criteria:

* Subject with a CL/P of known etiology,
* Subject with a NSCL/P and an IRF6 mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic factors | Day 1
  Identification of genetic factors implicated in orofacial cleft using whole exome sequencing (WES).

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte DEMEER, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens Picardie, Amiens, France